CLINICAL TRIAL: NCT05052437
Title: Open, Multicenter, Phase Ic Clinical Study on the Pharmacokinetics and Drug Interactions of Utidelone Plus Capecitabine in Patients With Recurrent and Metastatic Breast Cancer
Brief Title: PK and Drug Interaction Study of Utidelone Plus Capecitabine in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Chengdu Biostar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BG01-2001
Record Dates: First submitted 2021-05-30; First posted 2021-09-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Advanced and Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Utidelone (Experimental)
  Interventions: Drug: Utidelone
- Utidelone plus capecitabine (Experimental)
  Interventions: Drug: Utidelone Injection; capecitabine

INTERVENTIONS:
Drug: Utidelone Injection; capecitabine — 8 patients will be assigned to utidelone plus capecitabine arm receiving utidelone plus capecitabine. Utidelone injection 30mg/m2/day, intravenously administered once a day for 5 consecutive days; capecitabine tablets, 1000mg/m2, orally, 2 times a day for 14 consecutive days. 21 days is a cycle
  Arms: Utidelone plus capecitabine
Drug: Utidelone — 8 patients will be assigned to utidelone arm and receive utidelone injection 30 mg/m2/day intravenously, once a day for 5 consecutive days in a 21-day cycle.
  Arms: Utidelone

SUMMARY:
This trial is an open, multi-center, phase Ic clinical study on the pharmacokinetics and drug interactions of utidelone injection combined with capecitabine in patients with recurrent and metastatic breast cancer.

The purpose of this trial is:

1. To evaluate the pharmacokinetic characteristics of continuous intravenous administration of utidelone.
2. To evaluate the drug interaction of utidelone and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form, have good compliance, and cooperate with relevant inspections.
2. Histologically and/or cytologically diagnosed patients with advanced, metastatic breast cancer.
3. Patients who have previously received at least one anthracycline and taxane drug therapy (neoadjuvant therapy, adjuvant therapy, or recurrence and metastasis therapy), or the investigator believes that they can be included in this study.
4. Age ≥18 years; physical condition score ECOG 0~2 points.
5. Within 4 weeks before enrollment, Neuropathy should be less than grade 2 (NCI CTCAE 5.0).
6. Within 1 week before enrollment, routine blood examinations were basically normal (based on the normal value of each research center laboratory):

   1. White blood cell count (WBC) ≥3.0×109/L;
   2. Neutrophil count (ANC) ≥ 1.5×109/L;
   3. Platelet count (PLT) ≥100×109/L.
   4. Hemoglobin ≥9g/dL.
7. Within 1 week before enrollment, liver and kidney function tests were basically normal (the normal value of each research center laboratory is standard):

   1. Total bilirubin (TBIL)≤1.5×upper limit of normal (ULN);
   2. Alanine aminotransferase (SGPT/ALT)≤2.5×ULN (for liver metastases≤5×ULN);
   3. Aspartate aminotransferase (SGOT/AST)≤2.5×ULN (for liver metastases≤5×ULN);
   4. Creatinine clearance rate (Ccr) ≥60 ml/min.
8. No major organ dysfunction.
9. The patient must agree to provide blood, urine and stool samples for pharmacokinetic studies, and collect them in strict accordance with the required time points and intervals.
10. No mental abnormality, able to understand and undertake informed consent.

Exclusion Criteria:

1. Those who need to receive non-investigative anti-cancer therapy (such as chemotherapy, immunotherapy or biological therapy) during the administration period of this trial.
2. People who are severely allergic to castor oil, or who have had serious adverse reactions to anti-microtubule drugs in the past.
3. Within 4 weeks before receiving treatment, have had any major surgery or suffered major trauma; or are expected to undergo major surgery during the treatment.
4. Pregnancy (positive pregnancy test), breastfeeding patients, or those who are unwilling to use contraception during the test;
5. Those with uncontrollable intracranial hypertension syndrome (persistent headache, short-term blurred vision, and/or diplopia)
6. Combined serious diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, severe infection, active peptic ulcer, etc.
7. Known HIV infection, or untreated active hepatitis B or C;
8. Known to have alcohol or drug addiction, or have a history of uncontrollable mental illness, lack of legal capacity or limited legal capacity;
9. The investigator believes that it is inappropriate to participate in this trial.
10. Participate in another clinical trial or use other research treatments at the same time.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 12 weeks
  To measure the maximal plasma concentration of the study drugs and evaluate the pharmacokinetic characteristics of continuous intravenous administration of utidelone, measure PK parameters such as Maximum Plasma Concentration [Cmax]
C-T curve | 12 weeks
  To evaluate the pharmacokinetic interaction of utidelone and capecitabine in patients when administered in combination.
Area under the plasma concentration versus time curve (AUC) | 12 weeks
  To get area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
Measure and plot r-t curve | 12 weeks
  To analyse mass balance
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
  To evaluate the safety of the study

CONTACTS AND LOCATIONS:
Overall Officials: Quchang Ouyang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No